CLINICAL TRIAL: NCT03427515
Title: Effect of Supplementation With Saccharomyces Boulardii and Lactobacillus Rhamnosus on Examination-related Stress in Healthy Medical Students: a Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Probiotics and Examination-related Stress in Healthy Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Michal Karbownik, Research assistant, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 502-03/5-108-03/502-54-157
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Healthy; Stress-related Problem; Anxiety
Keywords: Psychobiotics; Probiotics; Examination; Stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Healthy medical students were assigned
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactobacillus (Experimental): Lactobacillus rhamnosus GG (ATCC 53103) - encapsulated
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG (ATCC 53103)
- Placebo (Placebo Comparator): Placebo - encapsulated mixture of maltodextrins
  Interventions: Dietary Supplement: Placebo
- Saccharomyces (Experimental): Saccharomyces boulardii (CNCM I-1079) - encapsulated
  Interventions: Dietary Supplement: Saccharomyces boulardii (CNCM I-1079)

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG (ATCC 53103) — 30 days of supplementation, 6x10^9 CFU/day
  Arms: Lactobacillus
Dietary Supplement: Saccharomyces boulardii (CNCM I-1079) — 30 days of supplementation, 5x10^9 CFU/day
  Arms: Saccharomyces
Dietary Supplement: Placebo — 30 days of supplementation
  Arms: Placebo

SUMMARY:
Probiotics are live microorganisms exhibiting multiple properties beneficial to health. An increasing body of evidence indicates that probiotics may support healthy brain function and may relieve stress. Recent research in this area has examined lactic acid bacteria in detail, but little is known about the stress-relieving effects of Saccharomyces, a yeast with probiotic properties.

Psychological stress is a factor that allows people to successfully cope with various daily life situations. On the other hand, excessive stress may lead to bodily harm and decrease performance, e.g. academic achievements. Probiotics may help manage stress, but little is known whether probiotics improve performance under stress.

The aim of this trial is to examine whether the healthy medical students may demonstrate better performance in academic examinations when supplementing their diet with a yeast probiotic strain Saccharomyces boulardii (CNCM I-1079) or bacterial probiotic strain Lactobacillus rhamnosus GG (ATCC 53103). The secondary aim of the trial is to evaluate the potential effects of this supplementation on state anxiety as well as on biochemical and physiological stress markers.

ELIGIBILITY:
Inclusion Criteria:

* Being a third year medical student of the Faculty of Medicine or Faculty of Military Medicine, Medical University of Lodz

Exclusion Criteria:

* formal inability to sit the first attempt of the final examination of Basic Medical Pharmacology
* chronic diseases: neurological, psychiatric, cardiological, gastroenterological, immunological, endocrine or infectious
* state of immunosuppression
* history of hospitalization (< 3 months before entrance to the study)
* presence of central venous catheter
* parenteral nutrition
* current pregnancy or intention to become pregnant within 3 months from the entrance to the study
* current lactation
* allergic reaction (< 3 months before entrance to the study)
* hypersensitivity to yeast, maltodextrins, potato starch, magnesium stearate, hypromellose, gelatin, glycerol or titanium dioxide
* body mass index over 30
* chronic medication use (current or < 3 months before entrance to the study)
* systemic antibacterial or antifungal medication use (current or < 3 months before entrance to the study)
* overuse of alcohol or psychoactive substances (current or < 3 months before entrance to the study)
* tobacco smoking - more than 5 cigarettes (or equivalents) a day (currently or < 3 months before entrance to the study)
* pro- or prebiotic preparations intake (< 3 months before entrance to the study)
* vegan or other atypical diet
* doing professional or extreme sports

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2016-06-20 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
Performance under examination-related stress | The examination is held on the 30th day of the trial.
  Number of correctly-answered questions in the final examination in Basic Medical Pharmacology

SECONDARY OUTCOMES:
State anxiety under examination-related stress | 30 minutes before the final examination in Basic Medical Pharmacology
  State anxiety measured with State-Trait Anxiety Inventory (STAI)
Cortisol | Measured a day before the final examination in Basic Medical Pharmacology
  Salivary cortisol level
Pulse rate | 30 minutes before the final examination in Basic Medical Pharmacology
  Individual, instructed measurement of pulse rate
Metanephrine | Measured a day before the final examination in Basic Medical Pharmacology
  Salivary metanephrine level

CONTACTS AND LOCATIONS:
Overall Officials: Michał S. Karbownik, PhD, Principal Investigator — Medical University of Lodz

REFERENCES:
- [Background] Dinan TG, Stilling RM, Stanton C, Cryan JF. Collective unconscious: how gut microbes shape human behavior. J Psychiatr Res. 2015 Apr;63:1-9. doi: 10.1016/j.jpsychires.2015.02.021. Epub 2015 Mar 3. PMID 25772005
- [Background] Foster JA, Rinaman L, Cryan JF. Stress & the gut-brain axis: Regulation by the microbiome. Neurobiol Stress. 2017 Mar 19;7:124-136. doi: 10.1016/j.ynstr.2017.03.001. eCollection 2017 Dec. PMID 29276734
- [Background] McFarland LV. Systematic review and meta-analysis of Saccharomyces boulardii in adult patients. World J Gastroenterol. 2010 May 14;16(18):2202-22. doi: 10.3748/wjg.v16.i18.2202. PMID 20458757
- [Derived] Karbownik MS, Kreczynska J, Kwarta P, Cybula M, Wiktorowska-Owczarek A, Kowalczyk E, Pietras T, Szemraj J. Effect of Supplementation with Saccharomyces Boulardii on Academic Examination Performance and Related Stress in Healthy Medical Students: A Randomized, Double-Blind, Placebo-Controlled Trial. Nutrients. 2020 May 19;12(5):1469. doi: 10.3390/nu12051469. PMID 32438624